CLINICAL TRIAL: NCT03069443
Title: Isometric Handgrip Home Training to Lower Blood Pressure in Hypertensive Older adulTs: a 20-week Assessor-blindEd raNdomized Controlled Trial
Brief Title: Isometric Handgrip Home Training to Lower Blood Pressure in Hypertensive Older adulTs
Acronym: POTENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Odense University Hospital (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Martin Joergensen, Senior researcher, cand. scient., PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POTENT
Record Dates: First submitted 2017-01-13; First posted 2017-03-03 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
Keywords: Isometric handgrip training; home training; older adults; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHG+Hypertension lifestyle guidelines (Experimental): Participants in this group will follow a home-based IHG training protocol. The IHG training will be structured with four sets of 2-minute contractions for each hand, 3 days per week for 20 weeks. In addition, the IHG group will receive information about hypertension-guidelines on lifestyle changes.
  Interventions: Other: IHG home training
- Hypertension lifestyle guidelines (No Intervention): The usual care group will receive information about hypertension-guidelines on lifestyle changes. The usual care group will have the same amount of hospital visits for measurements of blood pressure and maximal muscle tests as the intervention group in order to ensure similar attention provided by the healthcare professionals.

INTERVENTIONS:
Other: IHG home training — Participants of the intervention group will follow the IHG home training protocol for 20 weeks. The IHG training consists of isometric contractions applied with the hands on a Wii.
  Arms: IHG+Hypertension lifestyle guidelines

SUMMARY:
This Study evaluates the effect of 20 weeks of isometric handgrip (IHG) home training in adults aged 50 years or more. Half of the participants will serve as a control group and will only receive hypertension-guidelines on lifestyle changes.

DETAILED DESCRIPTION:
Hypertension markedly increases the risk of cardiovascular diseases and overall mortality. Lifestyle modifications such as increased levels of physical activity are recommended as the ﬁrst line of anti-hypertensive treatment. A recent systematic review showed that isometric handgrip (IHG) training was superior to traditional endurance and strength training in lowering resting systolic blood pressure (SBP). The average length of previous IHG training studies is approximately 7.5 weeks with the longest being 10 weeks. Therefore, presently it is unknown if it is possible to further lower blood pressure levels beyond the 10 week mark. Recently, the investigators developed a novel method for monitoring handgrip intensity using a standard Nintendo Wii Board (Wii). The primary aim of this study is to explore the effects of 20-weeks IHG home training facilitated by a Wii in hypertensive older adults (+50 years of age) in lowering SBP compared to usual care. Secondary aims are to explore if/when a leveling off effect on SBP will occur during the 20-week intervention period in the training group and to explore adherence and potential harms related to the IHG home training.

Methods: Based on previous evidence, the investigators calculated that 50 hypertensive older adults (+50 years of age) is needed to achieve a power of 80% or more. Participants will be randomly assigned to either an intervention group (IHG home training + hypertension-guidelines on lifestyle changes) or to a control group (hypertension-guidelines on lifestyle changes). Participants in the intervention group will perform IHG home training (30% of maximum grip strength for a total of 8 min per day per hand) three times a week for 20-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age +50 years old
2. Un-medicated (anti-hypertensive medicine) with resting SBP between 135-179 mmHg or hypertensive patient medicated with no change in treatment for ≥ 4 months with resting SBP between 135-179 mmHg

Exclusion Criteria:

1. Manifest cardiovascular disease (cerebrovascular disease, Heart failure, Chronic Kidney Disease, peripheral vascular disease, and advanced retinopathy (fundus hypertonus III-IV)).
2. Diabetes (any type)
3. More than three blood pressure regulating agents
4. Physical limitation preventing IHG training (e.g. missing an arm or musculoskeletal disorders).
5. Arthritis in the hand or carpal tunnel
6. SBP ≥ 180 mmHg (will be advised to see a doctor)

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | after 20 weeks of training
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)

SECONDARY OUTCOMES:
Diastolic blood pressure | after 20 weeks of training
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)
heart rate | after 20 weeks of training
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)
Handgrip maximum strength | baseline, 5 week, 15 weeks, and 20 weeks followup
  This will be measured using the WII and reported in kilograms in the FysioMeter software
Handgrip Rate of force development | baseline, 5 week, 15 weeks, and 20 weeks followup
  measured using a specially designed software working together with a standard wii board.
Handgrip Force variability | after 20 weeks of training
  This will be a measure of the muscle force variability during the isometric training sessions throughout the study
Visual Analog Pain Scale (VAS) | after 20 weeks of training
  At the end of each training session. Pain will be assessed for each hand/side using the VAS scale
Compliance to training sessions | after 20 weeks of training
  A report will be generated on how many sessions each participant have completed during the study
Systolic blood pressure | week 25, 35, and 40 post-intervention
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)
Diastolic blood pressure | week 25, 35, and 40 post-intervention
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)
heart rate | week 25, 35, and 40 post-intervention
  measured using a standard hospital electrical sphygmomanometer (Omron Comfort M6 AC)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University hospital, Aalborg, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data from the study will be made available on a public server

REFERENCES:
- [Derived] Jorgensen MG, Ryg J, Danielsen MB, Madeleine P, Andersen S. Twenty weeks of isometric handgrip home training to lower blood pressure in hypertensive older adults: a study protocol for a randomized controlled trial. Trials. 2018 Feb 9;19(1):97. doi: 10.1186/s13063-018-2441-x. PMID 29426359